CLINICAL TRIAL: NCT07243119
Title: PRIMA-HF PRedicting Recovery of Left Ventricular Function With Multimodality Cardiac IMAging in Patients With de Novo Heart Failure HAI-HF: High-Dose Adenosine During Perfusion Imaging in Heart Failure: Rationale and Design of the HAI-HF Trial
Brief Title: PRIMA-HF: Predicting Myocardial Recovery in Heart Failure Using Cardiac Imaging HAI-HF: High Dosing vs. Standard Dosing Adenosine During Myocardial Perfusion in Heart Failure
Acronym: PRIMA-HF
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Principal Investigator, Sarah Lindhøj Kvorning, Principal Investigator, MD, PhD student, Gødstrup Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1-10-72-126-25
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure and Reduced Ejection Fraction; Heart Failure
Keywords: LVEF; HFrEF; HFrecEF; Perfusion Imaging; Adenosine; Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose then High-dose Adenosine (Experimental)
  Interventions: Diagnostic Test: HAI-HF: Adenosine Stress [¹⁵O]H₂O PET Imaging; Drug: Two different doses of adenosine
- High-dose then Low-dose Adenosine (Experimental)
  Interventions: Diagnostic Test: HAI-HF: Adenosine Stress [¹⁵O]H₂O PET Imaging; Drug: Two different doses of adenosine

INTERVENTIONS:
Diagnostic Test: HAI-HF: Adenosine Stress [¹⁵O]H₂O PET Imaging — HAI-HF: Patients will be randomized in a 1:1 ratio to one of two dosing sequences: high-dose followed by low-dose adenosine, or low-dose followed by high-dose adenosine.
Drug: Two different doses of adenosine — Testing if high dose adenosine (210 ug/kg/min) during perfusion imaging results in a higher myocardial blood flow compared to standard dose (140 ug/kg/min) in patients with HFrEF

SUMMARY:
Background:

Heart failure with reduced ejection fraction (HFrEF) is a heterogeneous condition with variable potential for left ventricular ejection fraction (LVEF) recovery. While LVEF improvement and reverse remodeling predict better outcomes, the determinants that predict left ventricular recovery remain poorly understood. An expert panel of the Journal of American College of Cardiology highlighted the need for improved HFrEF phenotyping to clarify recovery patterns and support personalized management and risk stratification.

Methods:

PRIMA-HF is a prospective prediction study designed to determine whether baseline cardiac multimodality imaging can predict LVEF recovery in patients with de novo HFrEF (n=180). The imaging protocol includes cardiac magnetic resonance (CMR), coronary computed tomography and [¹⁵O]H₂O positron emission tomography ([¹⁵O]H₂O-PET) and echocardiography. Patients will also undergo a six-minute walk test, blood volume measurement, and blood sampling. The primary outcome is the change in LVEF from baseline to approx. after 3-12 months (or after full optitration in GDMT), assessed by CMR.

In 60 patients from the PRIMA-HF cohort, the randomized, double-blind study High Dose Adenosine During Perfusion Imaging in Heart Failure (HAI-HF) will be conducted. HAI-HF evaluates whether high-dose adenosine (210 µg/kg/min) versus standard-dose (140 µg/kg/min) during [¹⁵O]H₂O-PET changes the stress myocardial blood flow, which is the primary endpoint.

Aim:

The PRIMA-HF study comprehensively characterizes patients with newly diagnosed HFrEF through multimodality imaging and systematically assesses change in LVEF using CMR. The study's deep phenotyping approach integrates clinical, imaging, biomarker, and functional data to capture disease heterogeneity, rather than relying on traditional measures such as LVEF or symptom class. This enables the identification of distinct patient subgroups with shared pathophysiological mechanisms.

The HAI-HF trial examines whether higher adenosine doses improve [¹⁵O]H₂O-PET perfusion imaging in HFrEF.

Together, the studies will advance understanding of myocardial recovery, improve perfusion assessment, and support development of a predictive model for HFrEF prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Capable and has provided written informed consent
* LVEF ≤ 40% by echocardiography in connection with hospitalization for heart failure or in connection with outpatient evaluation for heart failure

Exclusion Criteria:

* Previous diagnosis of heart failure
* Unable to understand the patient information
* Pregnancy, as the study involves ionizing radiation.
* Current severe valvular disease (as defined by the Danish national treatment guidelines on cardio.dk)
* Atrial fibrillation with a heart rate > 130 beats per minute during the inclusion echocardiography
* Cardiac surgery within 6 months prior to inclusion
* Acute exacerbation of existing chronic obstructive pulmonary disease
* Severe asthma or chronic obstructive pulmonary disease with FEV1 < 1L
* any contraindication for adenosine stress testing
* Severe renal failure < 15 mL/min/1.73m² or dialysis
* Advanced liver disease (Child-Pugh class C)
* Endocarditis at inclusion/baseline
* Isolated right-sided heart failure
* Malignant disease treated with chemotherapy or radiotherapy, or expected life expectancy under 1 year

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
PRIMA-HF: Left ventricular ejection fraction (LVEF) | PRIMA-HF: Baseline through study completion, an average of 3 months
  Change in LVEF (continuous variable, absolute change in LVEF in percent points)
HAI-HF: Stress Myocardial Blood Flow (MBF) | Baseline and periprocedural
  Change in stress MBF (continuous variable, ml/min/g)

SECONDARY OUTCOMES:
PRIMA-HF: Kansas City Cardiomyopathy Questionaire (KCCQ-12) | Baseline through study completion, an average of 3 months
  Change in Kansas City Cardiomyopathy Questionnaire (KCCQ-12) (points, continuous data)
PRIMA-HF: 6 minutes-walk-test | Baseline through study completion, an average of 3 months
  Change in 6MWT distance (meters, continuous data)

OTHER OUTCOMES:
PRIMA-HF: Blood volume | Baseline through study completion, an average of 3 months
  Change in blodvolume (L, continuous data)
PRIMA-HF: NT-Pro-BNP | Baseline through study completion, an average of 3 months
  Change in NT-Pro-BNP (pg/mL or pmol/L, continuous data)

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Cardiovascular Reseach, Herning, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The study will adhere to all applicable regulations and guidelines governing the transfer of individual participantdata (IPD), which will be biological material (blood samples), abroad, ensuring that all data are handled confidentially and in full compliance with relevant legislation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing is planned after the enrollment of 200 patients in PRIMA-HF, which is anticipated to be achieved by the end of 2027. Approximately two months thereafter, we expect to have completed the necessary analyses, at which point the availability of individual participant data will cease.
  Upon completion of the project, collaborating partners will destroy all data in accordance with our agreements and applicable requirements.
Access Criteria: We plan to send biological material for proteomics measurements for further analysis to either deCODE, Reykjavik, Iceland, or Olink, Uppsala, Sweden. This will only take place after legal approval has been obtained in the Central Denmark Region.

REFERENCES:
- [Background] Funaya H, Kitakaze M, Node K, Minamino T, Komamura K, Hori M. Plasma adenosine levels increase in patients with chronic heart failure. Circulation. 1997 Mar 18;95(6):1363-5. doi: 10.1161/01.cir.95.6.1363. PMID 9118500
- [Background] Kim IC, Yoo BS. Multidimensional Approach of Heart Failure Diagnosis and Prognostication Utilizing Cardiac Imaging with Biomarkers. Diagnostics (Basel). 2022 Jun 1;12(6):1366. doi: 10.3390/diagnostics12061366. PMID 35741176
- [Background] Wilcox J, Yancy CW. Stopping medication for heart failure with improved ejection fraction. Lancet. 2019 Jan 5;393(10166):8-10. doi: 10.1016/S0140-6736(18)32825-3. Epub 2018 Nov 11. No abstract available. PMID 30429051
- [Background] Wilcox JE, Fang JC, Margulies KB, Mann DL. Heart Failure With Recovered Left Ventricular Ejection Fraction: JACC Scientific Expert Panel. J Am Coll Cardiol. 2020 Aug 11;76(6):719-734. doi: 10.1016/j.jacc.2020.05.075. PMID 32762907
- [Background] Postnov DD, Tuchin VV, Sosnovtseva O. Estimation of vessel diameter and blood flow dynamics from laser speckle images. Biomed Opt Express. 2016 Jun 22;7(7):2759-68. doi: 10.1364/BOE.7.002759. eCollection 2016 Jul 1. PMID 27446704
- [Background] Borges JP, Lopes GO, Verri V, Coelho MP, Nascimento PM, Kopiler DA, Tibirica E. A novel effective method for the assessment of microvascular function in male patients with coronary artery disease: a pilot study using laser speckle contrast imaging. Braz J Med Biol Res. 2016 Sep 1;49(10):e5541. doi: 10.1590/1414-431X20165541. PMID 27599202
- [Background] Strobeck JE, Feldschuh J, Miller WL. Heart Failure Outcomes With Volume-Guided Management. JACC Heart Fail. 2018 Nov;6(11):940-948. doi: 10.1016/j.jchf.2018.06.017. Epub 2018 Oct 10. PMID 30316941
- [Background] Bello D, Shah DJ, Farah GM, Di Luzio S, Parker M, Johnson MR, Cotts WG, Klocke FJ, Bonow RO, Judd RM, Gheorghiade M, Kim RJ. Gadolinium cardiovascular magnetic resonance predicts reversible myocardial dysfunction and remodeling in patients with heart failure undergoing beta-blocker therapy. Circulation. 2003 Oct 21;108(16):1945-53. doi: 10.1161/01.CIR.0000095029.57483.60. Epub 2003 Oct 13. PMID 14557364
- [Background] Dewey M, Siebes M, Kachelriess M, Kofoed KF, Maurovich-Horvat P, Nikolaou K, Bai W, Kofler A, Manka R, Kozerke S, Chiribiri A, Schaeffter T, Michallek F, Bengel F, Nekolla S, Knaapen P, Lubberink M, Senior R, Tang MX, Piek JJ, van de Hoef T, Martens J, Schreiber L; Quantitative Cardiac Imaging Study Group. Clinical quantitative cardiac imaging for the assessment of myocardial ischaemia. Nat Rev Cardiol. 2020 Jul;17(7):427-450. doi: 10.1038/s41569-020-0341-8. Epub 2020 Feb 24. PMID 32094693
- [Background] Tersalvi G, Beltrani V, Grubler MR, Molteni A, Cristoforetti Y, Pedrazzini G, Treglia G, Biasco L. Positron Emission Tomography in Heart Failure: From Pathophysiology to Clinical Application. J Cardiovasc Dev Dis. 2023 May 17;10(5):220. doi: 10.3390/jcdd10050220. PMID 37233187
- [Background] Graversen CB, Rasmussen LD, Sundboll J, Wurtz M, Kragholm KH, Bottcher M, Winther S. Cardiac computed tomography for rule-out of ischaemic heart disease in patients with new-onset heart failure. Eur Heart J Cardiovasc Imaging. 2025 Apr 30;26(5):794-801. doi: 10.1093/ehjci/jeaf090. PMID 40085773
- [Background] Burger PM, Savarese G, Tromp J, Adamson C, Jhund PS, Benson L, Hage C, Tay WT, Solomon SD, Packer M, Rossello X, McEvoy JW, De Bacquer D, Timmis A, Vardas P, Graham IM, Di Angelantonio E, Visseren FLJ, McMurray JJV, Lam CSP, Lund LH, Koudstaal S, Dorresteijn JAN, Mosterd A; European Society of Cardiology's Cardiovascular Risk Collaboration (ESC CRC). Personalized lifetime prediction of survival and treatment benefit in patients with heart failure with reduced ejection fraction: The LIFE-HF model. Eur J Heart Fail. 2023 Nov;25(11):1962-1975. doi: 10.1002/ejhf.3028. Epub 2023 Sep 18. PMID 37691140
- [Background] Perera D, Clayton T, O'Kane PD, Greenwood JP, Weerackody R, Ryan M, Morgan HP, Dodd M, Evans R, Canter R, Arnold S, Dixon LJ, Edwards RJ, De Silva K, Spratt JC, Conway D, Cotton J, McEntegart M, Chiribiri A, Saramago P, Gershlick A, Shah AM, Clark AL, Petrie MC; REVIVED-BCIS2 Investigators. Percutaneous Revascularization for Ischemic Left Ventricular Dysfunction. N Engl J Med. 2022 Oct 13;387(15):1351-1360. doi: 10.1056/NEJMoa2206606. Epub 2022 Aug 27. PMID 36027563
- [Background] Kjaerulff MLG, Tolbod LP, Pryds K, Nielsen R, Madsen S, Luong TV, Gormsen LC. Clinical use of [15O]H2O/[18F]FDG viability positron emission tomography does not reliably predict left ventricular ejection fraction improvement or survival after revascularization. Eur Heart J Cardiovasc Imaging. 2025 May 30;26(6):969-979. doi: 10.1093/ehjci/jeaf041. PMID 39901814
- [Background] Basuray A, French B, Ky B, Vorovich E, Olt C, Sweitzer NK, Cappola TP, Fang JC. Heart failure with recovered ejection fraction: clinical description, biomarkers, and outcomes. Circulation. 2014 Jun 10;129(23):2380-7. doi: 10.1161/CIRCULATIONAHA.113.006855. Epub 2014 May 5. PMID 24799515
- [Background] Punnoose LR, Givertz MM, Lewis EF, Pratibhu P, Stevenson LW, Desai AS. Heart failure with recovered ejection fraction: a distinct clinical entity. J Card Fail. 2011 Jul;17(7):527-32. doi: 10.1016/j.cardfail.2011.03.005. Epub 2011 May 6. PMID 21703523
- [Background] Swat SA, Cohen D, Shah SJ, Lloyd-Jones DM, Baldridge AS, Freed BH, Vorovich EE, Yancy CW, Jonnalagadda SR, Prenner S, Kim D, Wilcox JE. Baseline Longitudinal Strain Predicts Recovery of Left Ventricular Ejection Fraction in Hospitalized Patients With Nonischemic Cardiomyopathy. J Am Heart Assoc. 2018 Oct 16;7(20):e09841. doi: 10.1161/JAHA.118.009841. PMID 30371257
- [Background] Solomon SD, Anavekar N, Skali H, McMurray JJ, Swedberg K, Yusuf S, Granger CB, Michelson EL, Wang D, Pocock S, Pfeffer MA; Candesartan in Heart Failure Reduction in Mortality (CHARM) Investigators. Influence of ejection fraction on cardiovascular outcomes in a broad spectrum of heart failure patients. Circulation. 2005 Dec 13;112(24):3738-44. doi: 10.1161/CIRCULATIONAHA.105.561423. Epub 2005 Dec 5. PMID 16330684
- [Background] Solomon SD, Skali H, Anavekar NS, Bourgoun M, Barvik S, Ghali JK, Warnica JW, Khrakovskaya M, Arnold JM, Schwartz Y, Velazquez EJ, Califf RM, McMurray JV, Pfeffer MA. Changes in ventricular size and function in patients treated with valsartan, captopril, or both after myocardial infarction. Circulation. 2005 Jun 28;111(25):3411-9. doi: 10.1161/CIRCULATIONAHA.104.508093. Epub 2005 Jun 20. PMID 15967846
- [Background] St John Sutton M, Pfeffer MA, Moye L, Plappert T, Rouleau JL, Lamas G, Rouleau J, Parker JO, Arnold MO, Sussex B, Braunwald E. Cardiovascular death and left ventricular remodeling two years after myocardial infarction: baseline predictors and impact of long-term use of captopril: information from the Survival and Ventricular Enlargement (SAVE) trial. Circulation. 1997 Nov 18;96(10):3294-9. doi: 10.1161/01.cir.96.10.3294. PMID 9396419
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Bozkurt B, Coats AJS, Tsutsui H, Abdelhamid CM, Adamopoulos S, Albert N, Anker SD, Atherton J, Bohm M, Butler J, Drazner MH, Michael Felker G, Filippatos G, Fiuzat M, Fonarow GC, Gomez-Mesa JE, Heidenreich P, Imamura T, Jankowska EA, Januzzi J, Khazanie P, Kinugawa K, Lam CSP, Matsue Y, Metra M, Ohtani T, Francesco Piepoli M, Ponikowski P, Rosano GMC, Sakata Y, Seferovic P, Starling RC, Teerlink JR, Vardeny O, Yamamoto K, Yancy C, Zhang J, Zieroth S. Universal definition and classification of heart failure: a report of the Heart Failure Society of America, Heart Failure Association of the European Society of Cardiology, Japanese Heart Failure Society and Writing Committee of the Universal Definition of Heart Failure: Endorsed by the Canadian Heart Failure Society, Heart Failure Association of India, Cardiac Society of Australia and New Zealand, and Chinese Heart Failure Association. Eur J Heart Fail. 2021 Mar;23(3):352-380. doi: 10.1002/ejhf.2115. Epub 2021 Mar 3. PMID 33605000
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992